CLINICAL TRIAL: NCT02154776
Title: A Phase 1 Dose Escalation Study of LEE011 in Combination With Buparlisib and Letrozole for the Treatment of HR+, HER2-negative Post-menopausal Women With Locally Advanced or Metastatic Breast Cancer.
Brief Title: Dose Escalation Study of LEE011 in Combination With Buparlisib and Letrozole in HR+, HER2-negative Post-menopausal Women With Advanced Breast Cancer.
Acronym: LeeBLet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLEE011A2112C
Record Dates: First submitted 2014-05-28; First posted 2014-06-03 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2018-07

CONDITIONS: Advanced or Metastatic Breast Cancer
Keywords: LEE011,; buparlisib,; letrozole,; HR +,; HER2 - negative,; post-menopausal,; breast cancer,; CDK 4/6,; PI3K,; MTD
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; NVP-BKM120; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LEE011 + buparlisib + letrozole (Experimental): open label, dose escalation evaluating max tolerated dose of the triple combination
  Interventions: Drug: LEE011; Drug: Buparlisib; Drug: Letrozole

INTERVENTIONS:
Drug: LEE011 — 3 weeks on and 1 week off
Drug: Buparlisib — daily
Drug: Letrozole — 2.5 mg daily;

SUMMARY:
This is a multi-center, open-label, non-randomized, phase I study

ELIGIBILITY:
Inclusion Criteria:

1. Women with advanced (recurrent or metastatic) breast cancer who received no prior therapy for advanced disease.
2. Patient is postmenopausal.
3. Patient may have received ≤ 2 lines of chemotherapy for metastatic or recurrent breast cancer in the dose-escalation phase.
4. Patient has a histologically and/or cytologically confirmed diagnosis of estrogen-receptor positive and/or progesterone receptor positive breast cancer by local laboratory.
5. Patient has HER2-negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test is required by local laboratory testing.
6. Patient must have either:

   * Measurable disease, i.e., at least one measurable lesion as per RECIST 1.1 criteria or at least one predominantly lytic bone lesion

Exclusion Criteria:

1. Patient who received any CDK4/6 or PI3K inhibitor.
2. Patient has active cardiac disease or a history of cardiac dysfunction including any of the following:

   * History of angina pectoris, symptomatic pericarditis, or myocardial infarction within 12 months prior to study entry
   * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
   * Documented cardiomyopathy
   * Patient has a Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO)
   * History of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality in the previous 12 months.
   * On screening, any of the following cardiac parameters: bradycardia (heart rate < 50 at rest), tachycardia (heart rate > 90 at rest), PR interval > 220 msec, QRS interval >109 msec, or QTcF >450 msec.

   Systolic blood pressure >160 or <90 mmHg
3. Patient is currently receiving any of the following medications:

   * That are known strong inducers or inhibitors of CYP3A4.
   * That have a known risk to prolong the QT interval or induce Torsades de Pointes.
   * That have a narrow therapeutic window and are predominantly metabolized through CYP3A4.
4. Certain scores on an anxiety and depression mood questionnaires

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-06-27 (Actual); Primary Completion 2016-10-26 (Actual); Study Completion 2016-10-26 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | 28 days
  Dose Escalation Phase: Frequency of DLTs at each dose level associated with administration of LEE011, buparlisib, and letrozole in a 28 day cycle
Safety and tolerability of the combination of LEE011, buparlisib, and letrozole | approximately 25 months
  Dose Expansion Phase: Incidence of AEs, SAEs (overal and severity), laboratory abnormalities, ECG, vital, dose interteruptions, dose reductions, and dose intensity as a measure of safety and tolerability.

SECONDARY OUTCOMES:
Safety and tolerabiity of the combination of LEE011, buparlisib, and letrozole | approximately 25 months
  Dose Escalation Phase: Incidence of AEs, SAEs (overall and severity), laboratory abnormalities, ECG, vital, dose interterruptions, dose reductions, and dose intensity as a measure of safety and tolerability.
Pharmacokinetic paramters such as AUClast and Cmax of LEE011, buparlisib, and letrozole in order to characterize the PK profiles | approximately 25 months
  Dose Escalation Phase: When given in combination as well any other clinically significant metabolites that may be identified
Pharmacokinetic paramters such as AUClast and Cmax of LEE011, buparlisib, and letrozole in order to characterize the PK profiles | approximately 25 months
  Dose Expansion Phase: When given in combination as well as any other clinically significant metabolites that may be identified
Disease control rate | approximately 25 months
  Dose Expansion Phase: Proportion of patients with the best overall response of CR (complete response), PR (partial response), or SD (stable disease)
PFS (progression free survival) | approximately 25 months
  Dose Expansion Phase: Time from date of start of treatment to date of first documented progression or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (5):
  - University of California at Los Angeles UCLA SC, Los Angeles, California
  - Horizon Oncology Center SC, Lafayette, Indiana
  - Medical University of South Carolina SC, Charleston, South Carolina
  - South Texas Accelerated Research Therapeutics SC, San Antonio, Texas
  - University of Utah / Huntsman Cancer Institute SC-3, Salt Lake City, Utah
- Novartis Investigative Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CLEE011A2112C can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=16810